CLINICAL TRIAL: NCT05892783
Title: Effect of Plantar Fascia Release on Patients With Chronic Non-Specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Essraa Mahmoud Abdel Aziz Farag, Essraa Mahmoud, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF release in CNSLB
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Intervention Model Description: two parallel arms interventional studies
Masking Description: due to the nature of the study, neither the participants nor the investigator will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): This group will receive myofascial release on the PF of both legs, namely foam rolling, plantar fascia specific stretching and soft tissue mobilization.
  Interventions: Other: manual treatment
- control group (No Intervention): This group will receive advice only.

INTERVENTIONS:
Other: manual treatment — soft tissue mobilization applied by the therapist on the plantar fascia of both legs and self massage and stretching using foam roller and self stretching.
  Arms: experimental group

SUMMARY:
The purpose of the current study is to determine the effect of myofascial release of plantar fascia on pain, back function, lumbar flexibility and pain pressure threshold for patients with CNSLBP.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a major cause of disability and represent a burden on healthcare services worldwide (Hong et al., 2013; Hoy et al., 2014). The prevalence suggested that approximately 540 million people have experienced 'activity-limiting' low back pain (LBP) for at least once in their lifetime (Hartvigsen et al., 2018).

Previous evidence suggested that all of those who experience LBP, about 30%-40% will continue experiencing symptoms beyond 3 months and thus, become chronic (Henschke et al., 2008; Traeger et al., 2014). Around 85% of those who experience any form of LBP have no precise diagnosis, therefore they are categorized as 'non-specific' LBP (Chou, 2010). Efforts have been done by the healthcare research to understand the mechanisms underlying the persistence of pain in chronic non-specific LBP (CNSLBP).

There are many factors that can cause LBP, although it is very difficult to determine the exact cause (Alemo & Sayadipour, 2008). Those factors may include genetic factors, aging, obesity, smoking, work-related factors such as heavy manual work and the prolonged sitting hours required in most of the jobs. Also psychosocial factors (such as monotonous work and low job satisfaction) and Physiological factors (such as inadequate trunk strength and low physical fitness) can cause LBP (Kumar et al., 2014; Wai et al., 2010a; Wai et al., 2010b; Shiri et al., 2010a; Shiri et al., 2010b).

The concept of regional interdependence is well-recognized in the field of physical therapy. It is well recognized that when there is a dysfunction in one anatomical region, adjacent regions can be affected, causing the patient to complain from these adjacent areas. This concept is well recognized in the phenomenon of referred or radiating pain (Wainner et al., 2007).

Previous studies found the necessity to find the correlations between these anatomical regions which can help us understand more the main reasons for a certain dysfunction and thus, find more effective treatments (Wainner et al., 2007). For example, Berglund et al. (2008), found a potential relationship between the thoracic spine and elbow impairments.

Several studies applied on rats, showed that the force generated by muscle fiber contraction is transmitted both longitudinally and laterally, via the intramuscular fascia to the surrounding muscles, tendons and the bones. That's why when myofascial release was applied on certain areas, adjacent joint were effected as in previous studies (Huijing & Jaspers, 2005).

Moreover, the structure and orientation of fascial fibers determine how force is transmitted through connective tissues to the surrounding elements (Stecco et al., 2013; Wilke et al., 2018). Recent data showed that in humans, the length of muscle fascicles is affected by the coupling between muscle and fascia (Karakuzu et al., 2017; Pamuk et al., 2016).

These anatomical correlations were investigated by several studies, which found intimate connections between muscles and other elements in the body by connective tissues called fascia, Myers called them fascial chains (Myers, 2020).

Treatments of fascial tissues became very popular in the musculoskeletal disorders (Engel et al., 2014; De las Pen˜as et al., 2005; Ndetan et al., 2012; Ong et al., 2004; Wardle et al., 2013). This is due to recent histologic findings and the discovery of contractile cells, free nerve endings, and mechanoreceptors which suggest that fascia plays a proprioceptive and mechanically active role (Schleip et al., 2019).

It was found that plantar fascia is connected to adjacent muscles through a myofascial chain, Myers called this the superficial back line (SBL). It expands from the plantar fascia (PF), over the Achilles tendon, the gastrocnemii muscles, the hamstrings, the sacrotuberous ligament, erector spinae muscles and, eventually, the epicranial fascia (Myers, 2020; Stecco et al., 2019; Wilke et al., 2016).

Previous reviews have shown that myofascial release (MFR) immediately increased range of motion of nearby joint or even distant joint along the same myofascial chain (Cheatham et al., 2015; Hughes & Ramer, 2019; Wiewelhove et al., 2019; Wilke et al., 2020; Wilke et al., 2020). This has also been investigated along the superficial back line (SBL) (Wilke et al., 2020).

This was investigated by several studies which found the correlation between the plantar fascia and lumbar spine. There was an acute increase in the ROM of the lower back of healthy volunteers, when myofascial release (MFR) such as single foam rolling was applied on the plantar surface (Grieve et al., 2015; Kwangsun et al., 2018). This implicate that fascial chains might be able to change their properties or functional capacities in non-adjacent areas along their course (Krause et al., 2016).

Many studies have been performed on applying myofascial release (MFR) on the SBL in healthy individuals but, unfortunately, there is a lack of knowledge on their efficacy on LBP and several musculoskeletal disorders. Since CNSLBP is affecting a great population, more studies are required to investigate the effect of MFR on the SBL in patients with CNSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Both genders between the age of 20-45 years old.
* BMI less than 30 Kg/m2.
* Patients diagnosed as CNSLBP (pain > 3 months).
* Minimum pain level 2 out of 10 in NPRS.
* Psychologically and mentally stable.
* At least on trigger point in the lumbar paraspinals.
* Minimal level of disability in ODI.
* Reduced hamstring flexibility.

Exclusion Criteria:

* Red flags (eg. Spinal fractures, tumors, infection).
* Cauda equina syndrome that requires urgent surgery.
* Pregnant patients.
* Previous lumbar surgery.
* Fibromyalgia.
* Disc lesions and spinal degenerative disease such as lumbar spondylosis.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain | Around 10 minutes
  Therapist will assess pain intensity by using the Arabic version of Pain Numerical Rating Scale. It is 10 cm horizontal line with zero marked on one end (representing no pain) and 10 marked on the other end (representing worst imaginable pain).The scale will be explained to the patients first, then they will be asked to mark the best value that locates their pain level.
Assessment of back function | Around 15 to 30 mins
  Back function will be assessed by using Oswestry disability index (ODI). The ODI is a functional scale that assesses the impact of LBP on daily activities. It is a self-administered, 10 item questionnaire in which: the first section rates the intensity of pain and the others describe its disability effect on typical daily activities.
  The patient will be asked to choose the answer that best describes his/her current functional status. If more than one statement is marked in each item, the highest score will be taken to give a total ODI score ranging from 0 to 50, which is multiplied by 2 to be expressed as a percentage score.
  The sum will be calculated and presented as a percentage, where 0% represents no disability and 100% represents the worst possible disability. Disability categorized within the scale as following: mild or no disability (0% -20%), moderate disability (21% -40%), severe disability (41% - 60%), incapacity (61% - 80%), restricted to bed (81% -100%).
Assessment of Lumbar flexibility | 15 to 30 mins
  Modified-Modified Schober's test. During lumbar flexion assessment, patients will be in the standing position, whereas the examiner will be in a kneeling position behind patients. The posterior superior iliac spines will be identified.
  A horizontal line will be made between both posterior superior iliac spines. One ink mark will be made at the level of the S2 vertebra, and another ink mark will be 15 cm above the first mark. The examiner will then fix a tape measure between those two marks. Next, the examiner will instruct the patient to bend forward. The new distance between the two marks will be measured. The change in the difference between the measurement marks in standing and in flexion will be used to specify the amount of lumbar flexion.
  Assessment of lumbar extension will be performed same way as for lumbar flexion with the exception that the examiner will instruct the patient to bend backward.
Assessment of trigger points | Around 30 mins
  Trigger points will be assessed by using pressure algometer. Diagnosing myofascial trigger points will be applied as follows:
  1. Tender spot in a taut band,
  2. Patient pain recognition on tender spot palpation,
  3. Predicted pain referral pattern (the pain distribution expected from a trigger point in that muscle), and
  4. Local twitch response (a transient local contraction of skeletal muscle fibers in response to palpation or needling)
Hamstring flexibility | 15 to 30 mins
  The hamstring flexibility will be measured using the passive straight leg raise test and a standard universal goniometer. The axis will be on the knee joint, the stationary arm will be parallel to the axis of the femur, and the movable arm parallel to the leg. With the knee held straight, the participant's leg will be moved passively into hip flexion until tightness is felt. At that point, the physical therapist will read the goniometer in degrees of motion. Three trials will be performed on each leg, and the average will be used for recorded.